CLINICAL TRIAL: NCT02501512
Title: Maturational Changes in Coordination of Breathing, Heart Rate and Swallowing in Newborn Infants - a Single-centre Pilot Study
Brief Title: Maturational Changes in Newborn Infants
Status: Completed | Type: Observational
Sponsor: Sven Schulzke (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor-Investigator, Sven Schulzke, Director, Department of Neonatology, University Hospital, Basel, Switzerland
Organization: University Hospital, Basel, Switzerland (Other)
Other Study IDs: 2015136
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Immature Newborn; Abnormal Coordination
Keywords: transesophageal signal; swallowing; newborn
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to extract and discriminate the signals of respiration, heart rate and swallowing from a standard ECG and EMG signal obtained using a special neonatal gastric tube. These signals will be compared with the standard monitoring signals in the neonatal intensive care unit (NICU). Further, they will be used to search for objectively quantifiable maturational coordination processes of respiration, heart rate and swallowing. Lastly, this study aims to identify changes in ECG/EMG-signals as a result of external stimuli (e.g. nursing interventions) in the NICU.

DETAILED DESCRIPTION:
Coordination of respiration, heart rate and swallowing in preterm and term neonates has been subject of various studies in the past; its impeccable functioning is a key criterion to be fulfilled before infants are discharged home from the NICU. Whether coordination abilities depend only on gestational age and how they can be diagnosed objectively remains controversial. Also, the ideal time point of starting to introduce suck feeds and to challenge coordination of breathing and swallowing is unknown and largely remains a matter of trial and error with the risk of causing iatrogenic aspirations of milk if babies are not ready for suck feeds. Successful coordination of swallowing and breathing is generally considered as a higher neurological function and it does represent a mile stone in overall child development. Therefore, measurement of its level of functioning could have the potential to serve as a predictor for neurological outcome. However, it is yet unknown to what extent difficulties in preterm infants allow predictions concerning their neurological development and future outcome. One of the major reasons for these unsolved questions lies in the lack of diagnostic tools to objectively measure suck-swallow-breathing coordination with sufficient accuracy, which make a precise analysis of coordination patterns in preterm infants almost impossible. Considering the relevance of these questions, it seems important to develop tools to observe coordination of breathing, heart rate and swallowing in neonates with possibly greater accuracy.

In this single-centre pilot study 15 preterm infants of 32 to 42 weeks gestational age will be included. Transesophageal ECG and EMG signals will be measured using an Edi-gastric tube (Maquet, Getinge Group, Solna Sweden), a CE-certified neonatal gastric tube equipped with electrodes. Due to the proximity of the esophageal electrodes within the gastric tube to the heart and diaphragm, esophageal ECG and EMG signals can be acquired and are probably less susceptible to motion artefacts of the baby than the commonly used skin electrodes. This is well known from measurements in adults. Moreover, motion of esophageal electrodes due to peristalsis, respiration and cardiac motion superimposes the ECG as baseline wander and might be a surrogate for the coordination abilities of preterm infants.

Using these novel esophageal data this study's goal is to obtain objective data representing maturational patterns of breathing, heart rate, and swallowing in preterm infants. Possibly derived coordination patterns might help to guide nurses and clinicians to introduce suck feeds and to develop specific early intervention strategies. Furthermore, if the gastric tube-EMG proves to be accessible in real time, it could potentially replace standard monitoring tools that require the use of skin electrodes in the future. This would not only facilitate nursing and preserve skin integrity but also simplify bonding between the parents and their infants in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent by legal representatives as documented by signature
* Gestational age of 32 to 42 weeks
* Study start possible in the course of participant's 4th-10th day of life
* Presumed NICU stay ≥ 5 days from study start onwards
* Need for a gastric feeding tube for clinical reasons for ≥ 5 days from study start onwards

Exclusion Criteria:

* Major congenital malformations
* Circulatory instability (in need of therapy with vasoactive substances)
* Endotracheal ventilation
* Infant in extremis

Ages: 4 Days to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 15 infants hospitalized in the NICU of the University Children's Hospital Basel who were born between 32 and 42 weeks gestational age in the course of their first two weeks of life.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Respiratory rate determined by transoesophageal EMG | 5 consecutive days during first two weeks of life
Heart rate determined by transoesophageal ECG | 5 consecutive days during first two weeks of life
Swallowing act determined by transoesophageal EMG | 5 consecutive days during first two weeks of life

SECONDARY OUTCOMES:
Agreement of beat-to-beat heart rate (inter-beat-interval) obtained from EMG signals with corresponding values from NICU monitoring | 5 consecutive days during first two weeks of life
  To find out whether oesophageal data has the potential to replace standard NICU monitoring.
Change of average value of respiratory rate over the measurement period | 5 consecutive days during first two weeks of life
  To evaluate whether maturational changes in respiratory rate can be determined by EMG analyses
Change of average value of heart rate over the measurement period | 5 consecutive days during first two weeks of life
  To evaluate whether maturational changes in heart rate can be determined by EMG analyses

CONTACTS AND LOCATIONS:
Overall Officials: Sven Schulzke, Prof, Principal Investigator — University Children's Hospital Basel
Locations (1):
- University Children's Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No